CLINICAL TRIAL: NCT01408056
Title: The Efficacy of Timolol 0.5% Gel Forming Solution for the Treatment of Ulcerated Hemangiomas
Brief Title: Timolol Option for Ulcerated Hemangiomas (TOUCH Trial)
Acronym: TOUCH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty with recruitment
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Society for Pediatric Dermatology (Other)
Responsible Party: Principal Investigator, Albert Yan, Chief, Section of Pediatric Dermatology, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-007923
Record Dates: First submitted 2011-03-10; First posted 2011-08-03 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Infantile Hemangiomas
Keywords: Hemangioma; Infantile Hemangioma; Ulcerated Hemangioma; Timolol; Beta blocker; Vascular anomaly
MeSH Terms: conditions — Hemangioma; Hemangioma, Capillary; Vascular Malformations | interventions — Timolol; Mupirocin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol 0.5% Gel Forming Solution (GFS) (Experimental): Half of enrolled subjects will receive topical Timolol
  Interventions: Drug: Timolol 0.5% Gel Forming Solution (GFS)
- Mupirocin 2% ointment (Active Comparator): Half of enrolled subjects will receive Mupirocin
  Interventions: Drug: Mupirocin 2% Ointment

INTERVENTIONS:
Drug: Timolol 0.5% Gel Forming Solution (GFS) — Dose-based escalation schedule for topical application:
  4-8 kg: Day 0-7: 1 drop every other day; Day 7-14: 1 drop daily; Day 14 - Day 60: 1 drop twice per day
  8-12 kg: Day 07: 1 drop daily; Day 7-14: 1 drop twice per day; Day 14 - Day 60: 2 drops twice per day
  Other Names: Timolol 0.5% topical
  Arms: Timolol 0.5% Gel Forming Solution (GFS)
Drug: Mupirocin 2% Ointment — Topical application twice per day for 60 days
  Other Names: Mupirocin
  Arms: Mupirocin 2% ointment

SUMMARY:
The purpose of this study is to determine whether Timolol 0.5% Gel Forming Solution is safe and effective in promoting wound healing of infantile ulcerated hemangiomas compared with standard conservative management with topical antibiotic.

DETAILED DESCRIPTION:
Ulceration is the most common complication associated with infantile hemangiomas. Ulceration and the delay in wound healing places patients at risk for infection, bleeding, pain and permanent scarring. Currently, the care of ulcerated hemangiomas is extremely difficult and patients are often subject to multiple treatment modalities.

In the past two years, the leading advance in the treatment of hemangiomas has been the use of the non-selective, oral beta-blocker propranolol to arrest growth and promote involution of hemangiomas. Recent literature also suggests beta-blockers may have a role in helping ulcerated wounds re-epithelialize.

The use of a topical non-selective beta-blocker on isolated ulcerated hemangiomas may promote early healing and reduce the number of complications associated with ulceration. Investigation is needed to explore the safety and tolerability of applying a topical beta-blocker on an ulcerated hemangioma and whether topical beta-blockade may be more efficacious than conservative care with topical antibiotics.

In this study, infants will be randomized to either receive a topical antibiotic (topical mupirocin 2% ointment twice per day) or a topical beta-blocker (Timolol 0.5% Gel Forming Solution) according to a dose-escalation schedule. Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed. Photographs and safety and efficacy measurements will be taken at each visit to assess response to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Infants weighing between 4-12kg
* Infants with corrected gestational age 44 weeks - 8 months of age
* Infant with an ulcerated hemangioma
* Informed consent

Exclusion Criteria:

* Ulceration larger than 16cm2
* Ulcerated hemangioma with active bleeding or infection at time of enrollment
* Disease threatening hemangioma meeting criteria for oral propranolol
* Previous treatment with topical/oral corticosteroid or propranolol
* Medical history of congenital heart disease with decreased cardiac output, stroke/cerebral vasculopathy, active reactive airway disease or metabolic disorder
* History of an allergic reaction to Mupirocin or Timolol
* Currently taking medication that would interact with beta-blockers

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to Wound Re-epithelization | At 3 months

SECONDARY OUTCOMES:
Reduction in Ulcer Surface Area and Depth | At 3 months
Investigator's Global Evaluation of Disease | At 3 months
  A scoring system developed to measure clinical improvement of ulcerated hemangioma.
Timolol Serum Level | Measured at 1 month into therapy
Evaluate number of participants with changes in Glucose levels after drug is applied | Baseline, day 7, day 14
  Glucose monitoring will be performed for patients receiving Timolol 0.5% GFS before and 1 hour after drug is applied in clinic.
  Glucose values < 60 mg/dL will be considered significant.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.
Evaluate number of participants with evidence of changes in blood pressure following administration of Timolol 0.5% GFS | Baseline, day 7, day 14
  Blood pressure monitoring will be performed for patients receiving Timolol 0.5% GFS before and 1 hour after drug is applied in clinic.
  Blood pressure values < 3rd percentile (systolic or diastolic) will be considered significant for hypotension.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.
Pain scores (presence or absence) on the Wong-Baker faces scale | Baseline, day 7, day 14, 1 month, 2 months
  Investigators will question caregivers about common complications of ulcerated hemangiomas (pain, infection, bleeding) at each visit throughout the study. Pain will be assessed using the Wong-Baker faces scale.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.
Number of participants with presence or absence of Infection | Baseline, day 7, day 14, 1 month, 2 months
  Investigators will question caregivers about common complications of ulcerated hemangiomas (pain, infection, bleeding) at each visit throughout the study. Infection will be clinically assessed by presence of drainage or exudate, and/or culture positivity.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.
Number of participants with presence (or absence) of active bleeding | Baseline, day 7, day 14, 1 month, 2 months
  Investigators will question caregivers about common complications of ulcerated hemangiomas (pain, infection, bleeding) at each visit throughout the study. Infection will be clinically assessed by presence of active bleeding.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.
Evaluate number of participants with changes in Heart Rate after drug is applied | Baseline, day 7, day 14
  Glucose and vital sign monitoring will be performed for patients receiving Timolol 0.5% GFS before and 1 hour after drug is applied in clinic.
  Heart rate values < 3rd percentile will be considered significant and indicative of bradycardia.
  Subjects will be seen in clinic on day 7, day 14, 1 month and 2 months into therapy and 1 month after therapy is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Albert C. Yan, MD, Principal Investigator — Children's Hospital of Philadelphia, Chair of Pediatric Dermatology; Vikash S. Oza, MD, Principal Investigator — Children's Hospital of Philadelphia, Attending Physician; Patrick McMahon, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Pope E, Chakkittakandiyil A. Topical timolol gel for infantile hemangiomas: a pilot study. Arch Dermatol. 2010 May;146(5):564-5. doi: 10.1001/archdermatol.2010.67. No abstract available. PMID 20479314
- [Background] Sivamani RK, Pullar CE, Manabat-Hidalgo CG, Rocke DM, Carlsen RC, Greenhalgh DG, Isseroff RR. Stress-mediated increases in systemic and local epinephrine impair skin wound healing: potential new indication for beta blockers. PLoS Med. 2009 Jan 13;6(1):e12. doi: 10.1371/journal.pmed.1000012. PMID 19143471
- [Background] Sans V, de la Roque ED, Berge J, Grenier N, Boralevi F, Mazereeuw-Hautier J, Lipsker D, Dupuis E, Ezzedine K, Vergnes P, Taieb A, Leaute-Labreze C. Propranolol for severe infantile hemangiomas: follow-up report. Pediatrics. 2009 Sep;124(3):e423-31. doi: 10.1542/peds.2008-3458. Epub 2009 Aug 10. PMID 19706583
- [Background] Khunger N, Pahwa M. Dramatic response to topical timolol lotion of a large hemifacial infantile haemangioma associated with PHACE syndrome. Br J Dermatol. 2011 Apr;164(4):886-8. doi: 10.1111/j.1365-2133.2010.10177.x. No abstract available. PMID 21158749
- [Background] Chamlin SL, Haggstrom AN, Drolet BA, Baselga E, Frieden IJ, Garzon MC, Horii KA, Lucky AW, Metry DW, Newell B, Nopper AJ, Mancini AJ. Multicenter prospective study of ulcerated hemangiomas. J Pediatr. 2007 Dec;151(6):684-9, 689.e1. doi: 10.1016/j.jpeds.2007.04.055. Epub 2007 Aug 24. PMID 18035154